CLINICAL TRIAL: NCT03170401
Title: Protein-enhanced Enteral Nutrition and Metabolomics in Critically Ill Trauma and Surgical Patients
Brief Title: Supplemental Enteral Protein in Critical Illness
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Grant E. O'Keefe, Professor of Surgery, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00007918; 1R01GM127790-01A1 (NIH)
Record Dates: First submitted 2017-04-18; First posted 2017-05-31 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-05

CONDITIONS: Nutrition Disorder; Trauma; Critical Illness
MeSH Terms: conditions — Nutrition Disorders; Wounds and Injuries; Critical Illness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- no protein supplementation (Active Comparator): subjects receiving enteral nutrition without any protein supplementation
  Interventions: Other: Standard enteral nutrition
- protein supplementation (Experimental): subjects receiving enteral nutrition with additional protein supplementation
  Interventions: Dietary Supplement: Protein supplementation

INTERVENTIONS:
Dietary Supplement: Protein supplementation — enteral protein supplementation
  Arms: protein supplementation
Other: Standard enteral nutrition — Standard enteral nutrition.
  Arms: no protein supplementation

SUMMARY:
The aim of this study is too determine the effect of enteral protein supplementation on biochemical measures of inflammation and protein metabolism in critically ill surgical patients. The investigators will also collect data on important clinical outcomes, including infectious complications, duration of mechanical ventilation and other measures of recovery from critical illness.

Hypothesis: That early supplemental protein will increase serum concentrations of transthyretin at three weeks after the onset of illness or injury. Secondarily, the investigators will test whether supplementation, reduces infectious complications and increases ventilator-free days.

DETAILED DESCRIPTION:
Critically ill patients are frequently undernourished. The investigator's observations indicate that surgical and trauma patients who require artificial nutrition are likely to be markedly undernourished during the first week of critical illness, will often require intensive and costly support for organ failure, have prolonged stays in the intensive care unit and extended hospitalizations. Nitrogen deficits are typically greater and receive less attention than caloric deficits. In some respects, the focus on avoiding caloric deficits may have missed the mark. A broader consideration of nutrient needs, such as protein, is required. For instance, there are observational data supporting the notion that protein intake is at least as important as caloric intake in promoting recovery in critical illness. Only recently have national guidelines (ASPEN 2016) begun to specifically address protein requirements (1.5 - 2.0 g/kg/day). For a number of years, the approach to these critically ill patients has included weekly measurements of 24 hour urine nitrogen excretion in order to better understand the protein deficits that develop. Based upon physician preference, the investigators can then use enteral protein supplementation to match the urinary nitrogen excretion in order to achieve net "zero" nitrogen balance. With supplemental protein administration, physicians are able to reduce this deficit and in some cases, generate a positive nitrogen balance. However, there are no data to indicate that this approach (which is included as part of the 2016 ASPEN guidelines) improves clinical outcomes. The most obvious mechanism whereby supplemental protein may influence outcomes by providing more metabolic substrate for protein building. Feeding the gut likely creates a more anabolic environment and additional protein may facilitate anabolism. However, it is not known whether protein supplementation improves markers of anabolism and protein synthesis. In this study, the investigators will measure the anabolic effect of supplemental protein by following serum transthyretin concentrations as part of the standard clinical care.The investigators postulate that supplemental protein will attenuate the drop in comparison to no supplemental protein and will hasten the return to normal concentrations.

The proposed study will test whether early, and standardized protein supplementation: (1) Increases protein delivery during the first 2 weeks after injury, (2) increases serum transthyretin concentrations at 3 weeks after injury (3) increases ventilator-free days.

Study aims:

The aim of this study is to determine the effect of enteral protein supplementation on biochemical measures of protein metabolism in critically ill surgical patients. The investigators will also collect data on important clinical outcomes, including infectious complications, duration of mechanical ventilation and other measures of recovery from critical illness. However, this study will not enroll a sufficient number of subjects to adequately test for differences in these clinical end-points.

Hypothesis: That early supplemental protein will, increase serum concentrations of transthyretin at three weeks after injury. Secondarily, the investigators will test whether supplementation reduces infectious complications and increases ventilator-free days.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill adult trauma (blunt and penetrating) victims
* Other critically ill surgical patients
* enteral nutrition required during the first 96 hours after injury
* expected to require nutritional support for at least 1 week

Exclusion Criteria:

* Significant chronic organ failure,
* severe malnutrition pre-existing prior to ICU admission
* not expected to survive from their traumatic injuries.
* intestinal discontinuity
* short bowel syndrome
* bowel obstruction
* enterocutaneous fistula
* intestinal ischemia
* massive gastrointestinal hemorrhage
* inability to obtain enteral access.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grant O'Keefe, MD, Principal Investigator — University of Washington
Locations (1):
- Harborview Medical Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential study subjects included those admitted to the trauma and surgical intensive care services at Harborview Medical Center. Patients were screened by a member of the study team and were considered for inclusion if they were receiving mechanical ventilation expected to require ICU care for >7 days, deemed ready to start enteral nutritional support by the attending physician within 24 - 72 hours of admission, and had no contraindications to full enteral support.
Pre-assignment Details: No enrolled subjects were excluded prior to assignment to groups.
Groups:
- no Protein Supplementation: trauma subjects receiving enteral nutrition without any protein supplementation
- Protein Supplementation: trauma subjects receiving enteral nutrition with additional protein supplementation
  Protein supplementation: half the subjects will receive protein supplementation via enteral feedings and half will not receive the protein supplementation
Period: Study Subject Enrollment
Arm/Group | no Protein Supplementation | Protein Supplementation
Started | 256 | 244
Completed | 256 | 244
Not Completed | 0 | 0
Period: Follow up and Data Analysis
Arm/Group | no Protein Supplementation | Protein Supplementation
Started | 256 | 244
Completed | 256 | 244
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the primary outcome of serum transthyretin concentrations 129/256 participants in the no protein supplementation arm, and 122/244 participants in the protein supplementation arm had data available for analysis.
Groups:
- no Protein Supplementation: trauma and critically ill surgical patients receiving enteral nutrition without any protein supplementation
- Protein Supplementation: trauma and critically ill surgical patients receiving enteral nutrition with additional protein supplementation
- Total: Total of all reporting groups
Arm/Group | no Protein Supplementation | Protein Supplementation | Total
Number analyzed (Participants) | 256 | 244 | 500
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 49 [32 to 61] | 45 [30 to 59] | 47 [31 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 60 | 114
  Male | 202 | 184 | 386
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 27 | 53
  Not Hispanic or Latino | 224 | 210 | 434
  Unknown or Not Reported | 6 | 7 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 10 | 5 | 15
  Asian | 11 | 9 | 20
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 17 | 20 | 37
  White | 210 | 204 | 414
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 6 | 12
Region of Enrollment [Number; unit: participants]
  United States | 256 | 244 | 500

OUTCOME MEASURES:

1. Primary Outcome: Serum Concentrations of Transthyretin at 3 Weeks After Injury.
Description: Transthyretin is a circulating biomarker of nutritional status and protein synthesis.
Time Frame: 3 weeks after admission for injury
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | no Protein Supplementation | Protein Supplementation
Number analyzed (Participants) | 129 | 122
mg/dl | 18.1 (8.0) | 18.9 (8.5)

2. Secondary Outcome: Ventilator-free Days.
Description: Ventilator-free days will measured in the standard way and indicate the number of days a subject was alive and not receiving mechanical ventilation during the first 28 days.
Time Frame: Within 28 days following admission to hospital following injury.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | no Protein Supplementation | Protein Supplementation
Number analyzed (Participants) | 256 | 244
days | 15.0 (9.7) | 13.9 (9.8)

3. Secondary Outcome: Ventilator Associated Pneumonia.
Description: Pneumonia diagnosed while the patient is receiving mechanical ventilation as recorded in the institutional administrative trauma registry and ICU quality assurance database.
Time Frame: At any point during the hospitalization.
Measure: Count of Participants; unit: Participants
Arm/Group | no Protein Supplementation | Protein Supplementation
Number analyzed (Participants) | 256 | 244
Participants | 58 | 45

ADVERSE EVENTS:
Time Frame: Duration of hospitalization to a maximum of 1 year.
Arm/Group | no Protein Supplementation | Protein Supplementation
All-Cause Mortality (participants affected / at risk) | 34/256 | 36/244
Serious Adverse Events (participants affected / at risk) | 31/256 | 62/244
Other Adverse Events (participants affected / at risk) | 136/256 | 164/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | no Protein Supplementation (N=256) | Protein Supplementation (N=244)
Adjudicated aspiration (Respiratory, thoracic and mediastinal disorders) | 7 | 15 — When dual and blinded review of all episodes of hypoxemia or interruption of enteral nutrition were determined to be due to tracheal aspiration of gastric contents.
Reintubation (Respiratory, thoracic and mediastinal disorders) | 22 | 46 — Subject required endotracheal intubation following a planned extubation.
Gastrointestinal perforation (Gastrointestinal disorders) | 2 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | no Protein Supplementation (N=256) | Protein Supplementation (N=244)
Diarrhea (Gastrointestinal disorders) | 95 | 119
Abdominal distention (Gastrointestinal disorders) | 20 | 27
Emesis (Gastrointestinal disorders) | 21 | 18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-12-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT03170401/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-20): https://cdn.clinicaltrials.gov/large-docs/01/NCT03170401/SAP_001.pdf